CLINICAL TRIAL: NCT05581576
Title: Open Label Assessment of Pitolisant (Wakix) as Adjunct Therapy for Patients With Refractory Restless Legs Syndrome
Brief Title: Pitolisant in Refractory Restless Legs Syndrome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: William Ondo, MD (Other)
Collaborators: Harmony Biosciences Management, Inc. (Industry)
Responsible Party: Sponsor-Investigator, William Ondo, MD, Principal Investigator, The Methodist Hospital Research Institute
Organization: The Methodist Hospital Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00033508
Record Dates: First submitted 2022-09-01; First posted 2022-10-14 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Restless Legs Syndrome
Keywords: Refractory
MeSH Terms: conditions — Restless Legs Syndrome | interventions — pitolisant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Pitolisant (Wakix) (Experimental): Pitolisant will be titrated weekly until maximum dosage of 35.6 mg. Titration is dependent on subjects response.
  Interventions: Drug: Pitolisant

INTERVENTIONS:
Drug: Pitolisant — Pitolisant initial dose 8.9 mg, titrated depending on symptomatic response.
  Other Names: Wakix

SUMMARY:
This is an open-label trial in Restless Legs Syndrome (RLS) patients inadequately treated with standard therapy, defined by an IRLS score greater than 15. Investigators hypothesize that the study drug, Pitolisant (Wakix), may improve RLS symptoms.

DETAILED DESCRIPTION:
This is an open-label trial in RLS patients who have been inadequately treated with standard therapies, defined by an IRLS > 15. This trial consists of four study center visits (weeks 0, 4, 8, and 16) and four telephone visits (weeks 1, 3, 11, and a post safety phone call at week 17).

Subjects will titrate pitolisant for three weeks, starting with a dose of 8.9 mg at week 1, then increase to 17.8 mg at week 2, and a final increase to maximum dosage of 35.6 mg at week 3. If subjects are unable to tolerate the highest dose, they may reduce their dose to 17.8 mg. Titration of the drug will be monitored via telephone visits. During weeks 0-8, subjects will continue to take their current RLS medications. From week 8-16, subjects may either reduce or stop their other RLS medications as mutually agreed upon with investigator.

Several questionnaire assessments will be conducted throughout the study to monitor the subjects. Subjects will complete the International RLS Rating Scale (IRLS), Restless Legs Syndrome - 6 Scale (RLS-6), RLS Quality of Life Questionnaire (RLSQoL), Fatigue Severity Scale (FSS), Hamilton Depression Scale (HDS), Montreal Cognitive Assessment (MoCA), Epworth Sleepiness Scale (ESS), Clinical Global Impressions (CGI), and Clinical Global Impressions-Change (CGI-C).

ELIGIBILITY:
Inclusion Criteria:

* RLS diagnosed by standard criteria with an IRLS > 15 while taking at least 1 RLS medication
* Stable RLS medications for at least 2 weeks prior to study entry

Exclusion Criteria:

* MoCA < 24
* Concurrent untreated sleep disorders, not felt to be stable
* Subjects with any significant, unstable cardiovascular, liver, lung, renal, psychiatric, or neurological diseases (not including RLS)
* Intravenous iron within 4 weeks of study entry
* Breast feeding or pregnancy determined by urine pregnancy test in subjects where pregnancy is possible (pre-menopausal, sexually active women)
* Subjects with previous allergic reaction or lack of tolerability to Pitolisant

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2022-09-20 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
International RLS Rating Scale (IRLS) | At week 8
  This is a subjective scale to measure the severity of RLS within the past week.

SECONDARY OUTCOMES:
The Restless Legs Syndrome - 6 Scale (RLS-6) | Baseline, 4 weeks, 8 weeks, and 16 weeks
  This scale measures the severity of daytime versus nighttime RLS symptoms.
Restless Legs Syndrome Quality of Life Questionnaire (RLSQoL) | Baseline, 4 weeks, 8 weeks, and 16 weeks
  This scale assess the quality of life in RLS patients.
Fatigue Severity Scale (FSS) | Baseline, 4 weeks, 8 weeks, and 16 weeks
  This scale evaluates the impact of fatigue patients are experiencing.
Hamilton Depression Scale (HDS) | Baseline, 4 weeks, 8 weeks, and 16 weeks
  This scale assess symptoms of depression.
Montreal Cognitive Assessment (MoCA) | Baseline, 4 weeks, 8 weeks, and 16 weeks
  This assessment detects mild cognitive impairment.
Epworth Sleepiness Scale (ESS) | Baseline, 4 weeks, 8 weeks, and 16 weeks
  This is a subjective scale that measures a patient's sleepiness.
Clinical Global Impressions - Change | 1 week, 2 weeks, 4 weeks, 8 weeks, 11 weeks, 16 weeks, and 17 weeks
  This scale assess how much a patients illness has improved or worsened when compared to a baseline state from the beginning of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: William Ondo, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States